CLINICAL TRIAL: NCT05985564
Title: Retrospective Comparative Study on Imaging Between the Bochdalek Hernia and Congenital Diaphragmatic Eventration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, yan song, doctor, Children's Hospital of Chongqing Medical University
Other Study IDs: ysong
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Bochdalek hernia group
  Interventions: Other: imaging diagnosis
- the congenital diaphragmatic eventration group

INTERVENTIONS:
Other: imaging diagnosis — no intervention
  Groups: The Bochdalek hernia group

SUMMARY:
The imaging manifestations of diaphragmatic hernia and diaphragmatic distension were retrospectively analyzed and summarized, combined with the surgical findings, to summarize the differences in indirect signs of diaphragmatic hernia and diaphragmatic distension, so as to achieve the purpose of differential diagnosis.Research contents: (1) To summarize the characteristics of indirect imaging signs in patients with diaphragmatic hernia, to sum up the incidence of each sign, to find new signs and the prognosis of each sign; (2) Summarize the characteristics of indirect imaging signs in patients with diaphragmatic distension, summarize the incidence of each sign, and search for new signs and the prognosis of each sign; (3) To summarize the differences in indirect signs of diaphragmatic hernia and diaphragmatic distension, as well as the differences in their incidence, and combined with their surgical findings, to summarize their image identification points

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diaphragmatic hernia with surgical treatment
* Clinical diagnosis of congenital diaphragmatic eventration with surgical treatment

Exclusion Criteria:

* Diaphragmatic hernia or congenital diaphragmatic eventration without surgical treatment
* Diaphragmatic hernia or congenital diaphragmatic eventration without imaging examination

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The Bochdalek hernia and the congenital diaphragmatic eventration were included in the study. They had undergone surgical treatment.The imaging results and the surgical results were analysis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The position of the stomach | 1 day during the test
  The position of the stomach through imaging examination and operation
The position of the small intestine | 1 day during the test
  The position of the small intestine through imaging examination and operation

SECONDARY OUTCOMES:
The morphology of the small intestine | 1 day during the test
  The normal morphology, dilation and stenosis of the small intestine through imaging examination
The position of the colon | 1 day during the test
  The position of the colon through imaging examination and operation
The morphology of the colon | 1 day during the test
  The normal morphology, dilation and stenosis of the colon through imaging examination

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alamo L, Gudinchet F, Meuli R. Imaging findings in fetal diaphragmatic abnormalities. Pediatr Radiol. 2015 Dec;45(13):1887-900. doi: 10.1007/s00247-015-3418-5. Epub 2015 Aug 9. PMID 26255159
- [Background] Brown BP, Clark MT, Wise RL, Timsina LR, Reher TA, Vandewalle RJ, Brown JJ, Saenz ZM, Gray BW. A multifactorial severity score for left congenital diaphragmatic hernia in a high-risk population using fetal magnetic resonance imaging. Pediatr Radiol. 2019 Dec;49(13):1718-1725. doi: 10.1007/s00247-019-04478-2. Epub 2019 Aug 14. PMID 31414145
- [Background] Goodfellow T, Hyde I, Burge DM, Freeman NV. Congenital diaphragmatic hernia: the prognostic significance of the site of the stomach. Br J Radiol. 1987 Oct;60(718):993-5. doi: 10.1259/0007-1285-60-718-993. PMID 3676659